CLINICAL TRIAL: NCT02390167
Title: User Performance of the ONYX NEXT Blood Glucose Monitoring System
Brief Title: Evaluation of a Ascensia ONYX NEXT Investigational Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCA-PRO-2014-004-01
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2017-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Persons With Diabetes (Experimental): Untrained Subjects WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System).
  Interventions: Device: ONYX NEXT BGMS

INTERVENTIONS:
Device: ONYX NEXT BGMS — Untrained Persons WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick and palm blood (and study staff tested subject fingerstick blood) using the ONYX NEXT BGMS. All BG results were compared to reference method results obtained with subject capillary plasma. Also, study staff tested venous blood from subjects WITH Diabetes and BG results were compared to reference method results obtained from the subjects' venous plasma.

SUMMARY:
The purpose of this study was to determine if untrained subjects with diabetes and without diabetes could operate the Investigational Blood Glucose Monitoring System (BGMS) and obtain valid glucose results.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Pregnancy
* Physical, visual or neurological impairments that would make the person unable to perform testing with the BGM
* Previously participated in a blood glucose monitoring study using the ONYX NEXT or ONYX PLUS BGMS
* Working for a medical laboratory, hospital, or other clinical setting that involves training on or clinical use of blood glucose monitors
* Working for a competitive medical device company, or having an immediate family member who works for such a company
* A condition which, in the opinion of the investigator or designee, would put the person or study conduct at risk

General enrollment guidelines:

* At least 70% of subjects will be younger than age 65
* At least 10% (approximately 10-15%) of subjects will be naive users
* At least 20% of subjects with diabetes will have type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, FACP, Principal Investigator — AMCR Institute; Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research
Locations (2):
- United States (2):
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Persons With and Without Diabetes: Untrained Subjects WITH and WITHOUT Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System).
  The ONYX NEXT BGMS: Untrained Persons WITH and WITHOUT Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick and palm blood (and study staff tested subject fingerstick blood) using the ONYX NEXT BGMS. All BG results were compared to reference method results obtained with subject capillary plasma.
Period: Overall Study
Arm/Group | Persons With and Without Diabetes
Started | 376
With Diabetes | 333
Without Diabetes | 43
Completed | 375
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 376
Age, Continuous [Mean (Full Range); unit: years] | 52.1 [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202
  Male | 174
Race/Ethnicity, Customized [Number; unit: Number of responses]
  Hispanic/Latino | 50
  Not Hispanic or Latino | 321
  Ethnicity Unknown or Not Reported | 5
  American Indian or Alaska Native | 7
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 52
  White | 292
  Race Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 376

OUTCOME MEASURES:

1. Primary Outcome: Percent of Self-Test Fingerstick Blood Glucose (BG) Results (From Subjects WITH Diabetes) Within +/- 15mg/dL (<100mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Untrained subjects WITH Diabetes (332) self-tested fingerstick blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15 mg/dL (<100 mg/dL YSI capillary plasma) and +/- 15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 329 (332 with diabetes-3) Blood glucose results were analyzed. Three subjects did not obtain meter BG result after three attempts.
Measure: Number; unit: Percent of Results within 15mg/dL/15%
Groups:
- Persons With Diabetes: Untrained Subjects WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System).
  ONYX NEXT BGMS: Untrained Persons WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick blood using the ONYX NEXT BGMS. All BG results were compared to reference method results obtained with subject capillary plasma.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 329
Percent of Results within 15mg/dL/15% | 99.4

2. Secondary Outcome: Percent of Alternate Site Palm Blood Glucose (BG) Results (From Subjects WITH Diabetes) Within +/- 15mg/dL (<100mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Untrained subjects WITH Diabetes (332) self-tested Alternate Site (AST) palm blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15 mg/dL (<100 mg/dL YSI capillary plasma) and +/- 15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 318 (332 with diabetes -14) Blood glucose results were analyzed. Nine (9) subjects with low blood sugar did not attempt palm testing per protocol. Five (5) subjects had low blood sugar; their palm results were not evaluable per protocol.
Measure: Number; unit: Percent of Results within 15mg/dL/15%
Groups:
- Persons With Diabetes: Untrained Subjects WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System).
  ONYX NEXT BGMS: Untrained Persons WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System). Subjects tested capillary palm blood using the ONYX NEXT BGMS. All BG results were compared to reference method results obtained with subject capillary plasma.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 318
Percent of Results within 15mg/dL/15% | 97.2

3. Secondary Outcome: Percent of Subject Fingerstick Blood Glucose (BG) Results (From Subjects WITH Diabetes) Within +/- 15mg/dL (<100mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method When Tested by Study Staff
Description: Study staff tested subject (332 WITH diabetes) fingerstick blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15 mg/dL (<100 mg/dL YSI capillary plasma) and +/- 15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 332 Blood glucose results from subjects with diabetes were analyzed.
Measure: Number; unit: Percent of Results within 15mg/dL/15%
Groups:
- Persons With Diabetes: Untrained Subjects WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System).
  ONYX NEXT BGMS: Untrained Persons WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System). Study staff tested subject fingerstick blood) using the ONYX NEXT BGMS. All BG results were compared to reference method results obtained with subject capillary plasma.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 332
Percent of Results within 15mg/dL/15% | 99.7

4. Secondary Outcome: Percent of Venous Blood Glucose (BG) Results (From Subjects WITH Diabetes) Within +/- 15mg/dL (<100mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method When Tested by Study Staff
Description: Study staff tested venous blood of 332 subjects WITH diabetes using an Investigational Blood Glucose Monitoring System (BGMS). Venous BGMS results were compared with subject venous plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer venous plasma BG results were used to calculate the percent of BGMS results within +/- 15 mg/dL (<100 mg/dL YSI venous plasma) and +/- 15% (>=100 mg/dL YSI venous plasma).
Time Frame: 1 hour
Population: 330 (332-2) Blood glucose results were analyzed. Two (2) subjects had unsuccessful venipuncture attempts, so no venous results were obtained for them.
Measure: Number; unit: Percent of Results within 15mg/dL/15%
Groups:
- Persons With Diabetes: Untrained Subjects WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System).
  ONYX NEXT BGMS: Untrained Persons WITH Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System).
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 330
Percent of Results within 15mg/dL/15% | 100

5. Secondary Outcome: Percent of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 15% of Laboratory Glucose Method Across the Tested Glucose Range
Description: Untrained subjects WITH Diabetes (332) and WITHOUT Diabetes (43) self-tested fingerstick blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15% of the laboratory reference method across the entire tested YSI glucose range.
Time Frame: 1 hour
Population: 372 (375-3) Blood glucose results were analyzed. Three subjects did not obtain meter BG results after three attempts.
Measure: Number; unit: Percent of Results within 15%
Groups:
- Persons With and Without Diabetes: Untrained Subjects WITH and WITHOUT Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System).
  The ONYX NEXT BGMS: Untrained Persons WITH and WITHOUT Diabetes Use the ONYX NEXT BGMS (Blood Glucose Monitoring System).
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 372
Percent of Results within 15% | 99.5

6. Secondary Outcome: Percent of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 20% of Laboratory Glucose Method Across the Tested Glucose Range
Description: Untrained subjects WITH diabetes (332) and WITHOUT diabetes (43) self-tested Fingerstick blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 20% of the laboratory reference method across the entire tested YSI glucose range.
Time Frame: 1 hour
Population: 372 (375-3) Blood glucose results were analyzed. Three subjects did not contain meter BG results after three attempts.
Measure: Number; unit: Percent of Results within 20%
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 372
Percent of Results within 20% | 99.7

7. Secondary Outcome: Percent of Self-Test Alternate Site Palm Blood Glucose (BG) Results Within +/- 15% of Laboratory Glucose Method Across the Tested Glucose Range
Description: Untrained subjects WITH diabetes (332) and WITHOUT diabetes (43) self-tested AST palm blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15% of the laboratory reference method across the entire tested YSI glucose range.
Time Frame: 1 hour
Population: 361 (375-14) Blood glucose results were analyzed. Nine (9) subjects with low blood sugar did not attempt palm testing per protocol. Five (5) subjects had low blood sugar; their palm results were not evaluable per protocol.
Measure: Number; unit: Percent of Results within 15%
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 361
Percent of Results within 15% | 96.7

8. Secondary Outcome: Percent of Self-Test Alternate Site Palm Blood Glucose (BG) Results Within +/- 20% of Laboratory Glucose Method Across the Tested Glucose Range
Description: Untrained subjects WITH diabetes (332) and WITHOUT diabetes (43) self-tested AST palm blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 20% of the laboratory reference method across the entire tested YSI glucose range.
Time Frame: 1 hour
Population: as for outcome 7
Measure: Number; unit: Percent of Results within 20%
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 361
Percent of Results within 20% | 98.6

9. Secondary Outcome: Percent of Subject Fingerstick Blood Glucose (BG) Results Within +/- 15% of Laboratory Glucose Method When Tested By Study Staff
Description: Study staff tested subject (332 WITH and 43 WITHOUT diabetes) fingerstick blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15% of the laboratory method across the entire tested YSI glucose range.
Time Frame: 1 hour
Population: 375 Blood glucose results were analyzed.
Measure: Number; unit: Percent of Results within 15%
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 375
Percent of Results within 15% | 99.7

10. Secondary Outcome: Percent of Subject Fingerstick Blood Glucose (BG) Results Within +/- 20% of Laboratory Glucose Method When Tested By Study Staff
Description: Study staff tested subject (332 WITH and 43 WITHOUT diabetes) fingerstick blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 20% of the laboratory method across the entire tested YSI glucose range.
Time Frame: 1 hour
Population: 375 Blood glucose results were analyzed.
Measure: Number; unit: Percent of Results within 20%
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 375
Percent of Results within 20% | 100

11. Secondary Outcome: Percent of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 12.5mg/dL (<100mg/dL) and Within +/- 12.5% (>=100 mg/dL) of Laboratory Glucose Method
Description: Untrained subjects WITH Diabetes (332) self-tested fingerstick blood using an Investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 12.5 mg/dL (<100 mg/dL YSI capillary plasma) and +/- 12.5% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 329 (332-3) Blood glucose results were analyzed. Three subjects did not obtain meter BG result after three attempts.
Measure: Number; unit: Percent of Results within12.5mg/dL/12.5%
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 329
Percent of Results within12.5mg/dL/12.5% | 98.5

12. Secondary Outcome: Percent of Responses From Persons WITH Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements Regarding BGMS
Description: Staff obtained responses from persons WITH Diabetes (332) using short questionnaires to provide feedback on instructions for use and the basic operation of the BGMS. Subjects could respond 'Strongly Agree' or 'Agree' or are 'Neutral' or 'Disagree' or 'Strongly Disagree'.
Time Frame: 1 hour
Measure: Number; unit: Percent of Subjects who responded
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 332
Percent of Subjects who responded
  I find it easy to do a blood test with this meter. | 97.9
  The meter display was easy to see and read. | 98.2
  It was easy to understand my test results. | 99.7
  I like the overall meter design. | 97.3
  I find the meter easy to use. | 97.9
  Instructions (User Guide) were easy to understand. | 97.6
  Instructions clearly explain how to run a test. | 98.5
  Instructions clearly explain meter error messages. | 99.4

13. Secondary Outcome: Percent of Responses From Persons WITH and WITHOUT Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements Regarding BGMS
Description: Staff obtained responses from persons WITH and WITHOUT Diabetes using short questionnaires to provide feedback on instructions for use and the basic operation of the BGMS. Subjects could respond 'Strongly Agree' or 'Agree' or are 'Neutral' or 'Disagree' or 'Strongly Disagree'.
Time Frame: 1 hour
Measure: Number; unit: Percent of Subjects who responded
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 375
Percent of Subjects who responded
  I find it easy to do a blood test with this meter. | 98.1
  The meter display was easy to see and read. | 98.4
  It was easy to understand my test results. | 99.7
  I like the overall meter design. | 97.6
  I find the meter easy to use. | 98.1
  Instructions (User Guide) were easy to understand. | 97.6
  Instructions clearly explain how to run a test. | 98.7
  Instructions clearly explain meter error messages. | 99.2

14. Secondary Outcome: Percent of Responses From Persons WITH Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements Regarding Views/Behaviors Related to Self-Monitoring Blood Glucose
Description: Staff obtained responses from persons WITH Diabetes using short questionnaires to provide feedback on views and behaviors related to managing their diabetes. Subjects could respond 'Strongly Agree' or 'Agree' or are 'Neutral' or 'Disagree' or 'Strongly Disagree' or 'Choose Not to Answer'.
Time Frame: 1 hour
Measure: Number; unit: Percent of Subjects who responded
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 332
Percent of Subjects who responded
  Acc:important to help me talk w my HCP. | 100
  Acc:important to help w self-monitor satisfaction. | 99.70
  Acc:important to help w managing my diabetes. | 99.40
  Acc:important to help prevent low blood sugar | 99.69
  Acc:important to understand food/exercise effects. | 99.70
  Acc:help w using results to better control diabete | 99.40
  Acc:important to achieve greater peace of mind. | 99.09
  I prefer the meter I just used to my regular meter | 92.09
  I use my meter - my care provider gave it to me. | 85.27
  I use my current meter -my insurance covers strips | 85.62
  I use my current meter-I think it is most accurate | 84.09

15. Secondary Outcome: Percent of Self-Test Fingerstick Blood Glucose (BG) Results (From Subjects WITH and WITHOUT Diabetes) Within +/- 15 mg/dL (<75 mg/dL) and Within +/- 15% (>= 75 mg/dL) of Laboratory Glucose Method
Description: Untrained subject WITH and WITHOUT diabetes self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15 mg/dL (< 75 mg/dL YSI capillary plasma) and +/- 15% (>= 75 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 372 (375 - 3) Blood glucose results were analyzed. Three subjects did not obtain meter BG results after three attempts.
Measure: Number; unit: Percent of Results within 15mg/dL/15%
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 372
Percent of Results within 15mg/dL/15% | 99.7

16. Secondary Outcome: Percent of Self-Test Alternate Site Palm Blood Glucose (BG) Results (From Subjects WITH and WITHOUT Diabetes) Within +/- 15 mg/dL (<75 mg/dL) and Within +/- 15% (>= 75 mg/dL) of Laboratory Glucose Method
Description: Untrained subject WITH and WITHOUT diabetes self-tested Alternate Site (AST) palm blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15 mg/dL (< 75 mg/dL YSI capillary plasma) and +/- 15% (>= 75 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 366 (375-9) Blood glucose results were analyzed. Nine (9) subjects with low blood sugar did not attempt palm testing per protocol.
Measure: Number; unit: Percent of Results within 15mg/dL/15%
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 366
Percent of Results within 15mg/dL/15% | 97.0

ADVERSE EVENTS:
Arm/Group | Persons With and Without Diabetes
Serious Adverse Events (participants affected / at risk) | 0/375
Other Adverse Events (participants affected / at risk) | 8/375
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persons With and Without Diabetes (N=375)
Hypoglycemia (Endocrine disorders) | 8 (8) — Subjects with hypoglycemia (defined by site as BG level < 70 mg/dL) had diabetes and hypoglycemia was resolved at the visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days